CLINICAL TRIAL: NCT02656654
Title: Pilot Study to Evaluate the Efficacy of and the Tolerance to a Body Bandage to Maintain Fluid Balance in Patients With Severe Sepsis or in Septic Shock in an ICU
Brief Title: COrporeal Compression at the ONset of Severe Sepsis and Septic Shock
Acronym: COCOON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LARGE 2014
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Severe Sepsis or Septic Shock; Fluid Resuscitation
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Whole-body compression

SUMMARY:
Early and adequate fluid resuscitation (< 6 hours) in patients with circulatory failure is essential but may exacerbate oedema, which may itself: 1) aggravate pulmonary lesions and prolong mechanical ventilation, 2) aggravate organ failure and 3) increase mortality notably in patients with acute renal failure. Improving fluid balance is considered crucial in the management of patients in septic shock, but the efficacy of the measures currently proposed (diuretics associated or not with albumin and/or dialysis) is controversial. The investigators hypothesize that a whole-body compression using a body bandage could reduce capillary leakage and thus lead to faster restoration of a normal transmural pressure gradient in postcapillary venules and improve venous return.

This is the first study to evaluate mechanical compression using a body bandage to reduce oedema in septic shock.

To do this, a whole-body compression will be set up within the 12 hours following admission. Water balance will be monitored daily throughout the duration of the compression and vital status of patients will be search at 7 days, 28 days and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from a person of trust,
* Patients aged 18 years or over,
* Admitted to a Medical ICU for less than 24 hours,
* For severe sepsis or septic shock and requiring fluid resuscitation because of hypotension and/or persistent signs of circulatory shock,
* On mechanical ventilation with orotracheal intubation,

Exclusion Criteria:

* Person not covered by national health insurance
* Recent abdominal or pelvic surgery,
* Contra-indication for a body bandage (PAD, Compartment Syndrome, acute rhabdomyolysis, wounds),
* Pregnant women,
* Patients with severe sepsis or septic shock for more than 24 hours,
* Patients who are moribund or in whom death is probably imminent (within 24h),
* Patients who have given instructions not to be resuscitated,
* Patients under ward of court.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Fluid balance | At 7 days

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CH Chalon sur Saône, Chalon-sur-Saône
  - CHU de DIJON, Dijon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dargent A, Large A, Soudry-Faure A, Doise JM, Abdulmalak C, Jonval L, Andreu P, Roudaut JB, Prin S, Charles PE, Payen D, Quenot JP; COCOONs study group. Corporeal Compression at the Onset of Septic shock (COCOONs): a compression method to reduce fluid balance of septic shock patients. Sci Rep. 2019 Aug 9;9(1):11566. doi: 10.1038/s41598-019-47939-2. PMID 31399609